CLINICAL TRIAL: NCT05522582
Title: Safety and Efficacy of Oral Methotrexate Tablets Combined With Immunotherapy During Radiotherapy for Unresectable/Metastatic Solid Tumors: a Single-center, Prospective Study
Brief Title: Methotrexate Combined With Immunotherapy During Radiotherapy for Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yancheng First People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Geng, Clinical Professor, Yancheng First People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-K-099
Record Dates: First submitted 2022-08-28; First posted 2022-08-31 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors
Keywords: anti-PD-1 monoclonal antibody, radiotherapy, methotrexate
MeSH Terms: interventions — Methotrexate; spartalizumab; Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- methotrexate+anti-PD-1 antibody+radiotherapy (Experimental): Tablets with 5mg methotrexate are taken orally twice a week during radiotherapy. With anti-PD-1 monoclonal antibody, 200mg, Q3W.
  Interventions: Drug: Methotrexate tablets; Drug: Anti-PD-1 monoclonal antibody; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Methotrexate tablets — Tablets with 5mg methotrexate are taken orally twice a week during the whole course of radiotherapy
  Other Names: MTX
Drug: Anti-PD-1 monoclonal antibody — Anti-PD-1 monoclonal antibody 200mg is given intravenously every 3 weeks from the first day of radiotherapy until or after the end of treatment.
  Other Names: PD-1 inhibitors
Radiation: Radiotherapy — 6～15MV X-ray, 2Gy/time, 5times/week. The duration of radiotherapy depends on the target lesion.

SUMMARY:
Immune checkpoint inhibitors, such as programmed death 1 (PD-1) and programmed cell death-Ligand 1 (PD-L1), offer new approaches for systemic treatment of tumors, but clinical efficacy remains limited. Previous studies by our team have found that methotrexate can activate anti-tumor immunity. The discovery of a new effect of this drug will improve tumor response to immunotherapy and prognosis of patients.

DETAILED DESCRIPTION:
Malignant tumor is a systemic and complex disease that seriously endangers human health, surgery is the preferred treatment for solid tumors. Due to the extensive invasion and metastasis of advanced tumors, radiotherapy and chemotherapy are the main treatment options. However, the tolerance of tumor to chemoradiotherapy often leads to treatment failure and poor prognosis. Immunotherapy provides a new approach for the systemic treatment of tumors, but the clinical efficacy is still limited. Therefore, it is important to find effective drugs to improve the tumor response to radiotherapy and immunotherapy. Previous studies by our team have found that methotrexate can activate anti-tumor immunity. The discovery of a new effect of this drug will improve tumor response to immunotherapy and prognosis of patients. The objective of this clinical trial is to explore the efficacy and safety of methotrexate combined with immunotherapy and radiotherapy in patients with unresectable/recurrence solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have unresectable/ metastatic solid tumors;
2. ≥ 18 years old;
3. Life expectancy of at least 3 months;
4. Eastern Cooperative Oncology Group performance status 0-2;
5. Have at least one measurable lesion ≥ 1 cm as defined by response criteria;
6. Adequate organ function.

Exclusion Criteria:

1. Subjects with a history of autoimmune diseases or syndromes;
2. Serious uncontrolled medical disorders or active infections;
3. Women who are pregnant or breastfeeding;
4. Subjects have other factors that may cause them to terminate the study, such as other serious medical conditions (including mental illness) that require combined treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to 3 months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions)
Treatment-related adverse events (AEs) | Up to 6 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0

SECONDARY OUTCOMES:
Numbers of CD3+, CD4+ and CD8+T lymphocyte subsets in peripheral blood detected by flow cytometry | Approximately 2 months
  Laboratory tests for T-cell detection will be performed before and after treatment.
Levels of IL-6, TNF-α and IFN-γ in peripheral blood detected by flow cytometry | Approximately 2 months
  Peripheral blood will be collected before, during and after treatment for laboratory serum cytokine detection.
Progression-free Survival (PFS) per RECIST 1.1 | Up to 12 months
  PFS is defined as the time from enrollment to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 36 months
  OS is defined as the time from enrollment to death from any cause during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Geng, M.D., Study Director — Yancheng First People's Hospital
Locations (1):
- Yancheng First People's Hospital, Yancheng, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No